CLINICAL TRIAL: NCT01022086
Title: Assessment of Cardiotoxicity by Cardiac MRI Versus MUGA Scans in Breast Cancer Patients Receiving Trastuzumab: A Double-Blinded Prospective Observational Pilot Study
Brief Title: Assessment of Cardiotoxicity by Cardiac Magnetic Resonance (CMR) in Breast Cancer Patients Receiving Trastuzumab
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: Cardiac CMR
Record Dates: First submitted 2009-11-27; First posted 2009-12-01 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Stage I-IV Breast Cancer (Neo-adjuvant, Adjuvant, Locally Advanced and Metastatic)
Keywords: Breast Cancer; Cardiotoxicity; Trastuzumab; Cardiac MRI
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Cardiotoxicity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Mandatory: Troponin I/T and BNP will be assessed at each CMR time-point (and measured as per the institution's standard biochemistry laboratory commercial assay techniques.
  Optional: For consenting patients only, peripheral venous blood samples will be drawn at each CMR time-point. Each sample will be obtained with a tourniquet free technique, then undergo centrifugation to prevent platelet degranulation and enable platelet free serum to be obtained. Serum will then be separated and stored at -800C for subsequent analysis. TGF β1, amino terminal propeptide of procollagen type I (PINP) and type III (PIIINP) and the carboxyterminal telopeptide of collagen type 1 (CITP) will be measured by radioimmunoassay with commercially available kits. The intra-assay variations for determining PINP, PIINP, and CITP are 7%, 5%, and 8% respectively. CITP will be measured by ELISA according to the manufacturer's instructions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- early stage/adjuvant: Analyses will also be stratified according to the patient's stage of disease (i.e. early stage/adjuvant, locally advanced/neoadjuvant, and metastatic) and type of chemotherapy regimen (i.e. anthracycline-containing vs. non-anthracycline).
  Interventions: Procedure: Cardiac MRI; Biological: Biomarker Testing
- locally advanced/neoadjuvant: Analyses will also be stratified according to the patient's stage of disease (i.e. early stage/adjuvant, locally advanced/neoadjuvant, and metastatic) and type of chemotherapy regimen (i.e. anthracycline-containing vs. non-anthracycline).
  Interventions: Procedure: Cardiac MRI; Biological: Biomarker Testing
- metastatic: Analyses will also be stratified according to the patient's stage of disease (i.e. early stage/adjuvant, locally advanced/neoadjuvant, and metastatic) and type of chemotherapy regimen (i.e. anthracycline-containing vs. non-anthracycline).
  Interventions: Procedure: Cardiac MRI; Biological: Biomarker Testing
- anthracycline-containing: Analyses will also be stratified according to the patient's stage of disease (i.e. early stage/adjuvant, locally advanced/neoadjuvant, and metastatic) and type of chemotherapy regimen (i.e. anthracycline-containing vs. non-anthracycline).
  Interventions: Procedure: Cardiac MRI; Biological: Biomarker Testing
- non-anthracycline containing: Analyses will also be stratified according to the patient's stage of disease (i.e. early stage/adjuvant, locally advanced/neoadjuvant, and metastatic) and type of chemotherapy regimen (i.e. anthracycline-containing vs. non-anthracycline).
  Interventions: Procedure: Cardiac MRI; Biological: Biomarker Testing

INTERVENTIONS:
Procedure: Cardiac MRI — Cardiac magnetic resonance (CMR) imaging, otherwise called a cardiac (heart) MRI is a safe and standard clinical test that creates detailed images of your heart. It uses a computer to create images of your heart as it is beating, producing both still and moving pictures of your heart and major blood vessels. This test will allow the health professionals to obtain images of your beating heart and to look at the structure and function. Cardiac MRIs can help diagnose and evaluate a number of diseases conditions (such as heart failure, and heart valve disease) and will help doctors decide how to treat or manage patients who have heart problems.
Biological: Biomarker Testing — In addition to undergoing CMR imaging, patients will also have blood tests for two proteins, which serve as markers of heart injury and heart failure. These are called BNP and Troponin. These blood tests are currently used in clinical practice, but their precise role in monitoring heart function in cancer patients has not been well studied. Since the precise cause of Trastuzumab-induced heart damage is currently unknown, it is hoped that these two blood markers will provide valuable insights into how this happens.
  Peripheral venous blood samples will also be drawn at each CMR time-point. TGF β1, amino terminal propeptide of procollagen type I (PINP) and type III (PIIINP) and the carboxy-terminal telopeptide of collagen type 1 (CITP) will be measured by radioimmunoassay.

SUMMARY:
Herceptin has shown significant improvement in breast cancer therapy and improved survival of patients over-expressing the HER-2 protein by 50%. However, Herceptin has shown to negatively affect the heart, and frequent heart monitoring with multiple gated acquisition (MUGA) scans is required. MUGA scans use radiation and are not very accurate. This study will use cardiac magnetic resonance images (CMRs) to evaluate heart function and compare to MUGA scans in patients receiving Herceptin for early-stage breast cancer. In addition, novel biomarkers will also be assessed at the same time to help identify possible patients at risk for developing heart toxicities.

DETAILED DESCRIPTION:
Currently, serial MUGA scans are the imaging modality of choice for monitoring cardiotoxicity. However, MUGA scans only measure LVEF at the cost of ionizing radiation and considerable inter-study variability, and do not reliably detect cardiomyopathy. CMR is a highly accurate technique and represents a promising imaging alternative. Because CMR is now considered the gold standard for measuring LVEF and subclinical alterations in cardiac structure and function, it will be used in this prospective observational pilot study to determine its effectiveness for monitoring cardiotoxicity in patients receiving trastuzumab. Serial CMR will be compared to serial MUGA scans, as they are routinely used for LVEF monitoring with trastuzumab therapy, in standard practice. Cardiac biomarkers will also be measured in relation to CMR and MUGA scans. Furthermore, we will determine the long-term clinical and prognostic implications of trastuzumab-induced cardiotoxicity detected by these various methods.

This will be a double-blinded prospective observational pilot study of breast cancer patients with overexpression of HER2 on breast pathology (using either immunohistochemistry [IHC] and/or fluorescence in-situ hybridization [FISH]), who have never received trastuzumab before, who will be treated with trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Histologically confirmed diagnosis of invasive breast carcinoma
* Histologically confirmed HER2 overexpression using IHC and/or FISH and/or DISH
* Planned treatment with Trastuzumab or TDM-1
* Baseline LVEF >50% by MUGA (ECHOs or any other type of cardiac scanning may be done as part of standard clinical care, at the investigator's discretion; ECHOs cannot be done in place of MUGA scans)

Exclusion criteria:

* Previous treatment with trastuzumab or any other anti-HER2 agent (e.g. lapatinib, pertuzumab, etc.)
* Pre-existing symptomatic Heart Failure (NYHA Class III or IV)
* Recent acute coronary syndrome (myocardial infarction, unstable angina) within the last six months
* Recent coronary revascularization (percutaneous coronary intervention or coronary bypass surgery) within six months
* Permanent atrial fibrillation
* Inability to undergo MRI (shrapnel, metallic implants/clips, pacemaker or defibrillator)
* Currently pregnant and/or nursing
* Planned or current use of other targeted biological therapies that can potentially cause cardiotoxicity (i.e. bevacizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a double-blinded prospective observational pilot study of breast cancer patients with overexpression of HER2 on breast pathology (using either immunohistochemistry [IHC] and/or fluorescence in-situ hybridization [FISH]), who have never received trastuzumab before, who will be treated with chemotherapy (as per standard of care) and trastuzumab. Target recruitment number will be 50 patients over 18-24 months.
  Systemic therapy will include chemotherapy as dictated by Cancer Care Ontario's systemic therapy practice guidelines for stage I-IV (i.e. early stage, locally advanced and metastatic) breast cancer patients with HER2 overexpression.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To compare CMR with MUGA scans for determining LVEF and LV volumes in breast cancer patients treated with trastuzumab. | Five years

SECONDARY OUTCOMES:
To examine the association between changes in biomarker levels and changes in cardiac structure and function as measured by CMR in breast cancer patients receiving trastuzumab. | Five years

OTHER OUTCOMES:
To determine the long-term prognostic significance of reduced LVEF and myocardial injury detected by CMR and biomarkers in breast cancer patients treated with trastuzumab. | Five years

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Odette Cancer Centre/Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Gong IY, Ong G, Brezden-Masley C, Dhir V, Deva DP, Chan KKW, Graham JJ, Chow CM, Thavendiranathan P, Dai D, Ng MY, Barfett JJ, Connelly KA, Yan AT. Early diastolic strain rate measurements by cardiac MRI in breast cancer patients treated with trastuzumab: a longitudinal study. Int J Cardiovasc Imaging. 2019 Apr;35(4):653-662. doi: 10.1007/s10554-018-1482-2. Epub 2018 Nov 2. PMID 30390170
- [Derived] Barthur A, Brezden-Masley C, Connelly KA, Dhir V, Chan KK, Haq R, Kirpalani A, Barfett JJ, Jimenez-Juan L, Karur GR, Deva DP, Yan AT. Longitudinal assessment of right ventricular structure and function by cardiovascular magnetic resonance in breast cancer patients treated with trastuzumab: a prospective observational study. J Cardiovasc Magn Reson. 2017 Apr 10;19(1):44. doi: 10.1186/s12968-017-0356-4. PMID 28395671